CLINICAL TRIAL: NCT02562079
Title: Vasculopathy, Inflammation and Systemic Sclerosis: The Role of Endothelial Cell Activation and OX40/OX40L in Modulation of T Lymphocyte Activation
Brief Title: Vasculopathy, Inflammation and Systemic Sclerosis
Acronym: VISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2011/37
Record Dates: First submitted 2014-12-29; First posted 2015-09-29 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Systemic Sclerosis
Keywords: T lymphocyte; OX40/OX40L
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- subjects SSc diagnosed (Experimental)
  Interventions: Biological: Blood samples; Biological: Biopsy
- subjects Localised sclerosis diagnosed (Experimental)
  Interventions: Biological: Blood samples; Biological: Biopsy
- subjects Sc (Experimental)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — * biological features of the standard follow-up
  * 2 more blood tube for the biological collection (serum and PBMC)
Biological: Biopsy — Skin biopsies
  Arms: subjects Localised sclerosis diagnosed; subjects SSc diagnosed

SUMMARY:
It is a study of basic research with mechanistically objectives and including clinical biological samples.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare and severe disease characterised by a fibrotic process and an incompletely elucidate physiopathology. Several shared featured have been identified between SSc and another autoimmune disease, the systemic lupus erythematous (SLE) as an interferon-alpha signature, the role of platelets and the polymorphism of OX40 ligand (OX40L). In SLE, OX40L has been shown highly linked to the active form of the disease, was increased by the CD40L of platelets and induced the CD8 cytotoxicity while inhibiting the suppressive functions of regulator T lymphocytes. The third main factor of the SSc physiopathology apart from autoimmunity and fibrosis is the vasculopathy with an important role of endothelial cells (EC). They turned out to be half-professional antigen presenting cells and can modulate the adaptive immunity.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75.
* SSc diagnosed according to the American College of Rheumatology (ACR) criteria.
* With skin manifestations since less than 10 years.
* Localised sclerosis (LSc) diagnosed, morphea type.

Exclusion Criteria:

* Age inferior to 18 or upper than 75.
* Skin manifestations since more than 10 years.
* Haemostasis diseases (independent from treatments).
* Stem cell transplant.
* Immunosuppressive treatments in the last 6 months.
* Associate autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of OX40L expression in endothelial cells and skin biopsies. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service de Rhumatologie - Tripode - Hôpital Pellegrin, Bordeaux, Bordeaux, France